CLINICAL TRIAL: NCT01304680
Title: Evaluation of Fluid Resuscitation in Children With Cancer With Severe Sepsis / Septic Shock
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Grupo de Apoio ao Adolescente e a Crianca com Cancer (Other)
Responsible Party: Principal Investigator, Priscila de Biasi, MD, Grupo de Apoio ao Adolescente e a Crianca com Cancer
Other Study IDs: UTI/IOP 03/11; 0101/11 (Other: CEP UNIFESP)
Record Dates: First submitted 2011-02-24; First posted 2011-02-25 (Estimated); Last update posted 2012-11-29 (Estimated); Status verified 2012-11

CONDITIONS: Cancer; Septic Shock; Other Fluid Overload
MeSH Terms: conditions — Neoplasms; Shock, Septic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Retrospective study to evaluate the characteristics of patients and of fluid resuscitation during intensive care unit hospitalization of patients under septic chock.

ELIGIBILITY:
Inclusion Criteria:

* patients admitted between Jan/2009 and Dec/2010
* patients with septic chock diagnosis

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: pediatric patients admitted to intensive care unit with septic chock
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2011-01

CONTACTS AND LOCATIONS:
Locations (1):
- Grupo de Apoio ao Adolescente e a Criança com Cancer, São Paulo, São Paulo, Brazil